CLINICAL TRIAL: NCT03711344
Title: Improving Access to High Quality, Culturally Relevant Treatment for East Asian Canadian Youth in Ontario
Brief Title: Culturally Adapting CBT for East Asian Youth in Ontario
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: East Metro Youth Services (Other); Hong Fook Mental Health Association (Unknown); Ontario Centre of Excellence for Child and Youth Mental Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: innovation-1927
Record Dates: First submitted 2018-09-11; First posted 2018-10-18 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Anxiety; Depression
Keywords: Cognitive Behavioral Therapy; Cultural Adaptation; East Asian Youth
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: East Asian youth diagnosed with Anxiety and/or depression will be randomly assigned to either the experimental group (receives the cultural adapted version of cognitive behavioral therapy) or the control group (non-culturally adapted cognitive behavioral therapy). It is a randomized control trial design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally adapted Cognitive Behavioral therapy (Experimental): The experimental group will receive the culturally adapted version of cognitive behavioral therapy.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Non-adapted Cognitive Behavioral therapy (Active Comparator): The control group will receive the original (non-adapted) version of cognitive behavioral therapy.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The intervention will be administered by therapists working at community agencies who are experienced at providing Cognitive Behavioral Therapy.

SUMMARY:
This mixed methods study proposes a culturally adapted cognitive behavioural therapy (CA-CBT) model for an East Asian demographic in Canada. The client population of East Asian youth who have been diagnosed with anxiety and/or depression are the focus of the study. CBT has been proven as a very effective form of therapy, and when adapted can promote positive mental health outcomes for a growing and increasingly vulnerable population. Developing a culturally adapted version of CBT (CA-CBT) for this population adds a practical treatment that improves access to culturally relevant care.

DETAILED DESCRIPTION:
There is a major lack of culturally relevant mental health services for East Asian youth in Ontario and Canada. Beginning with a participatory/qualitative research approach, common themes amongst clients, caregivers, healthcare professionals, and community leaders, will divulge basic elements needed to develop a culturally adapted model of cognitive behavioural therapy. The information from the adapted model will be taught to participating psychologists who will deliver the therapy in a randomized control trial design, with feasibility testing of the intervention using a quantitative approach ensuing. Immediate guidelines will then be developed for use by therapists working with East Asian youth.

ELIGIBILITY:
Inclusion Criteria:

* Self identification as East Asian origin
* Between the ages of 12 to 21
* Diagnosed as having depression and/or anxiety

Exclusion Criteria:

* Have been affected by psychosis
* Have been affected by serious addiction
* Have been affected by cognitive impairment

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-09-18 (Estimated); Study Completion 2019-09-18 (Estimated)

PRIMARY OUTCOMES:
Severity levels of depression and anxiety rated by the Hospital Anxiety and Depression Scale (HADS). | 4 months.
  Severity levels of depression and anxiety will be rated pre- and post-intervention by the Hospital Anxiety and Depression Scale (HADS). The scale ranges from 0 to 21 for anxiety and 0 to 21 for depression. A score of 0 to 7 for depression and/or anxiety is considered a normal range. A score of 8 to 10 suggests the potential presence of depression and/or anxiety. A score of 11 or more suggests a likely presence of depression and/or anxiety.
Severity levels of depression and anxiety rated by the Bradford Somatic Inventory (BSI). | 4 months.
  Severity levels of depression and anxiety will be rated pre- and post-intervention by the Bradford Somatic Inventory (BSI). The Bradford Somatic Inventory uses "yes" or "no" questions relating to somatic symptoms of anxiety and/or depression. A "yes" response to a question equates to a somatic symptom linked to depression and/or anxiety. The maximum number of "yes" responses is 46 and the minimum is 0. A higher number of "yes" responses suggests a potential increase in the severity of depression and/or anxiety.

SECONDARY OUTCOMES:
Satisfaction of the culturally adapted Cognitive Behavioral Therapy assessed using the Verona Satisfaction Scale. | 4 months.
  Satisfaction will be measured using the Verona Satisfaction Scale. This scale measures patients satisfaction with health care services. The items are rated by 4 categories labelled: "strongly disagree", "disagree", "agree", and "strongly agree", on a scale of 1 to 4. A higher sub-scale/domain score indicates better satisfaction. All sub-scales are summed up to compute total/domain score. This scale will be used to identify the strengths and weaknesses of the therapy service and provide guidance for further development.

CONTACTS AND LOCATIONS:
Overall Officials: Farooq Naeem, M.D., Principal Investigator — Centre for Addiction and Mental Health; Myra Levy, M.A., Study Director — East Metro Youth Services
Locations (1):
- East Metro Youth Services, Scarborough Village, Ontario, Canada